CLINICAL TRIAL: NCT00970463
Title: Impact of Growth Hormone on Serum N-Terminal Pro-B-Type Natriuretic Peptide (NT-proBNP) and on Cardiac Function and Morphology Evaluated by Magnetic Resonance Imaging in Growth Hormone Deficiency and Acromegaly
Brief Title: Cardiac Function and Morphology Evaluated by Magnetic Resonance Imaging in Growth Hormone Deficiency and Acromegaly
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Mikkel Andreassen MD, Department of Endocrinology, Herlev Hospital, Herlev ringvej, 2730 Herlev, Denmark
Other Study IDs: KA-20060035
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Growth Hormone Deficiency; Cardiac Function
Keywords: The GH-system and cardiac function
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GH: Patients with GHD
- Pegvisomant and Somatostatin analogues: Acromegaly

SUMMARY:
To test the hypothesis that both lack and excess of growth hormone (GH) is associated with cardiac abnormalities. Cardiac function and morphology will be evaluated by MRI before and after treatment.

DETAILED DESCRIPTION:
It is an open prospective noninterventional clinical study. Treatment and follow-up will be according to usual guidelines, and will be unaffected by inclusion in the study. GHD patients will be treated with daily subcutaneous GH injections. Patients with acromegaly will be treated with either transsphenoidal surgery or by medical treatment with long acting somatostatin analogues, dopamine agonist, GH antagonist or combinations of these treatment modalities.

Patients will be examined by Cardiac MRI before treatment and after one year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Peak GH below 6.0 ng/mL during Pyridostigmine-GHRH test.
* Nadir GH above 0.4 ng/mL and elevated levels of IGF-I during oral glucose tolerance test

Exclusion Criteria:

* Contraindications for magnetic resonance scan

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GHD based on an insufficient stimulation of GH-secretion during Pyridostigmin-GHRH test.
  Patients with acromegaly based on an insufficient supression of GH-secretion during oral glucose tolerance test
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac function i relation to changes in the activity of the GH-axis

REFERENCES:
- [Derived] Andreassen M, Faber J, Kjaer A, Petersen CL, Kristensen LO. Cardiac function in growth hormone deficient patients before and after 1 year with replacement therapy: a magnetic resonance imaging study. Pituitary. 2011 Mar;14(1):1-10. doi: 10.1007/s11102-010-0250-7. PMID 20730514